CLINICAL TRIAL: NCT00019110
Title: VACCINE THERAPY AND DETECTION OF IMMUNOLOGIC RESPONSES WITH HUMAN PAPILLOMAVIRUS 16 E6 AND E7 PEPTIDES IN PATIENTS WITH METASTATIC OR LOCALLY ADVANCED CERVICAL CANCER
Brief Title: Vaccine Therapy in Treating Patients With Advanced or Recurrent Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064330; NCI-95-C-0154; NCI-T94-0134N; NCT00001441 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 1999-11

CONDITIONS: Anal Cancer; Cervical Cancer; Esophageal Cancer; Head and Neck Cancer; Penile Cancer; Vulvar Cancer
Keywords: stage IV anal cancer; recurrent anal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; stage IIIA anal cancer; stage IIIB anal cancer; recurrent esophageal cancer; stage III cervical cancer; stage IV cervical cancer; recurrent cervical cancer; stage III vulvar cancer; stage IVB vulvar cancer; recurrent vulvar cancer; stage III penile cancer; stage IV penile cancer; recurrent penile cancer; recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage III squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III verrucous carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage IV salivary gland cancer; stage III salivary gland cancer
MeSH Terms: conditions — Anus Neoplasms; Uterine Cervical Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms; Penile Neoplasms; Vulvar Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — oncogene protein E7, Human papillomavirus type 16; E6 protein, Human papillomavirus type 16

INTERVENTIONS:
Biological: human papillomavirus 16 E7 peptide
Biological: synthetic human papillomavirus 16 E6 peptide

SUMMARY:
RATIONALE: Vaccines made from certain human papillomaviruses may be able to help the body to kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of human papillomavirus vaccine therapy in treating patients who have advanced or recurrent cancer of the cervix, vagina, penis, anus, esophagus, or head and neck.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether endogenous cellular immunity to the viral oncoproteins human papilloma virus 16 (HPV16) E6 and E7 is present in patients with advanced or recurrent carcinoma of the cervix or other carcinomas that carry HPV16.
* Determine whether vaccination with antigen-presenting cells pulsed with synthetic peptide corresponding to the tumor's HPV16 E6 or E7 peptide can induce or boost patient cellular immunity to that particular peptide.
* Determine the type and characteristics of the cellular immunity generated in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the tumor response in patients treated with this regimen.
* Determine whether in vivo T cells generated specifically against HPV16 E6 or E7 peptide can be cloned and expanded in vitro against the corresponding peptide.

OUTLINE: Patients are stratified according to disease category as defined by the following:

* Stratum A: Stage III cervical cancer not previously treated with appropriate radiotherapy; stage IV or recurrent cervical cancer; or other advanced tumors that harbor human papilloma virus 16 (HPV16) such as anogenital, esophageal, or head and neck cancers.
* Stratum B: Stage III cervical cancer previously treated with standard therapy with no evidence of residual disease. Vaccination in this group is given as adjuvant therapy.

Patients are assigned to receive HPV E6 or E7 peptide by the principal investigator. Peripheral blood mononuclear cells (PBMC) (antigen presenting cells) are harvested and treated in vitro with sargramostim (GM-CSF) and pulsed with HPV16 E6 or E7. Patients receive vaccination with HPV16 E6 or E7 pulsed PBMC IV over 1-2 minutes during weeks 1, 3, 7, and 11 for a total of 4 vaccinations. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (CR) continue treatment for a maximum of 1 year past CR.

Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 40-46 patients (at least 28 patients for stratum A and 12 for stratum B) will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage III, IV, or recurrent carcinoma of the cervix or other tumor that carries human papilloma virus 16 (HPV16) such as other anogenital (vulvar, penile, and anal), esophageal, and head and neck cancers
* HLA-A2.1 positive
* Patients with tumors other than cervical cancer must have no other therapeutic options
* Fresh tissue or paraffin block available for HPV genome detection and typing (optional for cervical cancer)
* No history of CNS metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-1

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGPT no greater than 4 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart disease

Immunologic:

* No autoimmune disease, e.g.:

  * Systemic lupus erythematosus
  * Multiple sclerosis
  * Ankylosing spondylitis
  * HIV negative
* Responsive to 1 of the following skin test antigens:

  * Mumps Trichophyton
  * Candida Tetanus

Other:

* No active infection requiring antibiotics
* No weight loss greater than 20% within the past 6 months
* No other active malignancy except basal cell skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* At least 4 weeks since prior steroids and recovered

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* Recovered from the toxic effects of prior therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-11

CONTACTS AND LOCATIONS:
Overall Officials: Barry L. Gause, MD, Study Chair — National Cancer Institute (NCI)
Locations (6):
- United States (6):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Center for Cancer Research, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Morristown Memorial Hospital, Morristown, New Jersey
  - University of Texas Medical Branch, Galveston, Texas